CLINICAL TRIAL: NCT05664503
Title: The Effect of Mobile Health Education on Adaptation to Stoma, Self-efficacy, and Peristomal Skin Lesions: A Quasi-experimental Study
Brief Title: The Effect of Mobile Health Education on Adaptation to Stoma, Self-efficacy, and Peristomal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Eylem Togluk Yigitoglu, Asisst. Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulU 2022-07/12
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Nurse's Role; Patient Compliance; Peristomal Skin Complication; Self Efficacy
Keywords: ostomy adjustment; mobile application; self-efficacy; peristomal skin lesions; nursing
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study with a post-test control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Booklet (No Intervention): Control-Classical patient education before the operation, the patient is educated with the classical method brochure.
- STOMA-M (Experimental): Patients are educated with the mobil aplikasyon method.
  Interventions: Other: Assigned Interventions STOMA-M

INTERVENTIONS:
Other: Assigned Interventions STOMA-M — The training, which includes information on stoma care, maintenance of daily life activities, and complication management, was given to the patients in the experimental group via the STOMA-M.
  Arms: STOMA-M

SUMMARY:
To explore the effect of the Stoma Mobile application-based training method on the psychosocial adjustment, self-efficacy, and development of peristomal skin complications in individuals with a stoma.

Quasi-experimental study with a post-test control group. Patients who met the inclusion criteria were randomly selected. While the experimental group (n=30) received training with the Stoma Mobile application, the control group (n=30) received training with the booklet. Stoma compliance, self-efficacy level, and the presence of complications were compared in both groups in the first and third months after discharge.

H11: Individuals who receive stoma care training via STOMA-M will have a higher adaptation to stomas than individuals who receive stoma care training via a booklet.

H12: The SE levels of individuals who receive stoma care training via STOMA-M will be higher than those who receive stoma care training via a booklet.

H13: Peristomal skin complications of individuals who receive stoma care training via STOMA-M will be lower than those who receive stoma care training via a booklet.

The population of the study included patients who had a stoma for the first time, were in a university hospital in Istanbul between December 2020 and December 2021, and who were 18 years of age and older, literate, without any physical and psychological disabilities, able to use smartphones, and willing to participate in the study. Patients who were in the same room or underwent a urostomy were not included in the study.

The experimental group using the Stoma Health Mobile application had higher psychosocial adjustment and self-efficacy scores than the control group, and the peristomal skin lesion complication rate was lower than that of the control group. Social self-efficacy positively affects stoma compliance, and the Stoma Mobile application positively affects the level of social self-efficacy and adaptation of ostomates to the stoma

DETAILED DESCRIPTION:
Ostomates need to learn to cope with new self-care routines and emotional problems related to changes in body image and self-perception. This learning process is defined as psychosocial adjustment. Adaptation of the patient to the stoma after surgery is part of the process in which the patient re-coordinates the body, self, and external world. In addition to the follow-up process after surgical treatments, psychosocial adjustment is one of the most important factors that define SE and quality of life.

Bandura (1994) defines SE as the belief that people can effectively initiate the necessary activities and reach results in events related to their lives. In other words, SE is a dynamic cognitive process that expresses the confidence of individuals with a stoma in their own ability to be successful in stoma care. SE plays an important role in adapting to the stoma. Not only do individuals who can self-care better adapt to a stoma.

Structured education has an important place in the ability of ostomates to cope with these problems. This training is indispensable, as it helps ostomates cope with physical, psychological, and social difficulties. Face-to-face training given during hospitalization is a traditional and effective method designed to impart new information and self-care behavior. However, it has its limitations. This type of training is time-consuming, and retaining the given information is often difficult for patients, as they experience postoperative anxiety and pain. In addition, the number of ostomy and wound care nurses in Turkey is not sufficient. When ostomates experience a problem with their stoma, they may not be able to contact the ostomy nurse. Considering that stomas are usually applied to cancer patients, their general condition deteriorates due to chemotherapy and radiotherapy. For this reason, it is important that ostomates receive information on living with a stoma in their mobile environment, thus having such information accessible at any time through their smartphones.

The literature contains limited studies comparing the effects of face-to-face/booklet and mobile training on the adaptation, self-efficacy, and peristomal skin complications of ostomates. Accordingly, this study evaluated the effect of the mobile application and booklet training in the education of ostomates on the adaptation and skin complications of ostomates. Thus, the study examined the effect of using innovative, technology-based education approaches in the education of ostomates, offering a significant contribution to the literature and individual-centered care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Literate,
* Without any physical and psychological disabilities,
* Able to use smartphones
* Willing to participate in the study.

Exclusion Criteria:

* Patients who were in the same room or underwent a urostomy were not included in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Adjustment Scale for Individuals with Ostomy | Evaluation of the differences between scales score - The scale is filled in 2 times; After being discharged from the hospital the first months(1) and third months (2)
  It is a self-assessment scale consisting of 23 items developed by to determine the compliance of individuals with stoma. The scale, which is graded in a five-point Likert type, has four sub-dimensions. These four dimensions are anger, social adaptation, anxiety/worry and acceptance. While the lowest score on the scale is '0', the highest score is '92'

SECONDARY OUTCOMES:
Stoma Self-Efficacy Scale | Evaluation of the differences between scales score - The scale is filled in 2 times; After being discharged from the hospital the first months(1) and third months (2)
  The scale consists of 22 items. The scale, which is graded in a five-point Likert type, consists of two sub-dimensions. Sub-dimensions; Stoma Care is Self-Efficacy and Social Self-Efficac. The possible score on the scale ranges from 22 to 110. The higher the score, the better the level of self-efficacy

OTHER OUTCOMES:
Evaluation Tool for Peristomal Skin Lesions; SACS | Evaluation of the differences between scales score - The scale is filled in 2 times; After being discharged from the hospital the first months(1) and third months (2)
  The SACS; The five most common lesions in the SACS (L) are: hyperemic (L1: peristomal redness with intact skin), abrasive (L2: open lesion not extending to subcutaneous tissue; skin loss in partial thickness), ulcerative (L3: open lesion extending to subcutaneous tissue and under the skin; skin loss in full-thickness), ulcerative (L4: skin loss in full-thickness with dead tissue), and proliferative (L5: abnormal growth present; i.e., hyperplasia, granulomas, neoplasms) lesions.
  Five topographic (T) quadrants arranged clockwise around the stoma are used to record the location of the peristomal lesion: TI: Left upper peristomal quadrant (between 12-3 o'clock), TII: Left lower peristomal quadrant (between 3-6 o'clock), TIII: Right lower peristomal quadrant (between 6-9 o'clock), TIV: Right upper peristomal quadrant (between 9-12 o'clock), and TV: Refers to all peristomal quadrants.

CONTACTS AND LOCATIONS:
Locations (1):
- Eylem Toğluk Yiğitoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yigitoglu ET, Sendir M. Effect of a mobile patient education application on adjustment to stoma and development of peristomal skin lesions: a quasi-experimental study. Wound Manag Prev. 2021 Dec;67(12):30-40. PMID 35030542
- [Background] Yigitoglu, E. T., & Sendir, M. (2021a). Mobile Application in Stoma Care Education: Stoma-M. Journal of Education and Research in Nursing, 18 (2), 210-216. DOI: 10.5152/jern.2021.85688
- [Background] Karacay P, Togluk Yigitoglu E, Karadag A. The validity and reliability of the Stoma Self-Efficacy Scale: A methodological study. Int J Nurs Pract. 2020 Dec;26(6):e12840. doi: 10.1111/ijn.12840. Epub 2020 Apr 17. PMID 32301580
- [Background] Karadağ, A., Göçmen, Z. B., Korkut, H., & Çelik, B. (2011). Turkish adaptation of the adjustment scale for individuals with ostomy. National Journal of Surgery, 27(4), 206-211.
- [Background] Ay A, Bulut H. Assessing the Validity and Reliability of the Peristomal Skin Lesion Assessment Instrument Adapted for Use in Turkey. Ostomy Wound Manage. 2015 Aug;61(8):26-34. PMID 26291898
- [Background] Pate K, Powers K, Coffman MJ, Morton S. Improving Self-Efficacy of Patients With a New Ostomy With Written Education Materials: A Quality Improvement Project. J Perianesth Nurs. 2022 Oct;37(5):620-625. doi: 10.1016/j.jopan.2021.11.020. Epub 2022 Mar 5. PMID 35260298
- [Background] Wang QQ, Zhao J, Huo XR, Wu L, Yang LF, Li JY, Wang J. Effects of a home care mobile app on the outcomes of discharged patients with a stoma: A randomised controlled trial. J Clin Nurs. 2018 Oct;27(19-20):3592-3602. doi: 10.1111/jocn.14515. Epub 2018 Jul 10. PMID 29775491
- [Background] Seo HW. Effects of the frequency of ostomy management reinforcement education on self-care knowledge, self-efficacy, and ability of stoma appliance change among Korean hospitalised ostomates. Int Wound J. 2019 Mar;16 Suppl 1(Suppl 1):21-28. doi: 10.1111/iwj.13047. PMID 30793857
- [Background] Wound, Ostomy and Continence Nurses Society; Guideline Development Task Force. WOCN Society Clinical Guideline: Management of the Adult Patient With a Fecal or Urinary Ostomy-An Executive Summary. J Wound Ostomy Continence Nurs. 2018 Jan/Feb;45(1):50-58. doi: 10.1097/WON.0000000000000396. PMID 29300288
- [Background] Yaşar, Z., & Üstündağ, H. (2021). Determination of quality of life and self-efficacy levels of patients with stoma. Journal of Celal Bayar University Health Sciences Institute, 8(1), 107-115.
- [Background] Collado-Boira EJ, Machancoses FH, Folch-Ayora A, Salas-Medina P, Bernat-Adell MD, Bernalte-Marti V, Temprado-Albalat MD. Self-Care and Health-Related Quality of Life in Patients with Drainage Enterostomy: A Multicenter, Cross Sectional Study. Int J Environ Res Public Health. 2021 Mar 2;18(5):2443. doi: 10.3390/ijerph18052443. PMID 33801488
- [Background] Heidari-Beni F, Esmaeilian S, Yousefi F, Zarei MR, Farahani MA. Comparison of Face-to-Face Education and Multimedia Software Education on Adjustment of Patients With Intestinal Ostomy: A Randomized Controlled Trial. J Wound Ostomy Continence Nurs. 2022 Mar-Apr 01;49(2):152-157. doi: 10.1097/WON.0000000000000854. PMID 35255067